CLINICAL TRIAL: NCT01291680
Title: Assessment of Central Pain in the Peripartum Period
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jacob N Ablin MD, Tel Aviv Souraski Medical Center
Other Study IDs: 0033-10-TLV
Record Dates: First submitted 2011-02-02; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Pre - Delivery Pregnant Women; Chronic Pain; Pain During Delivery
Keywords: Pregnancy; Chronic pain; Fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre - delivery pregnant women: Participants in the study will be pregnant women attending the obstetric ER for routine term followup. This evaluation is generally conducted at week 39-41 of pregnancy. The current study will focus on women attending a regular followup, not considered to be at high risk.

SUMMARY:
Chronic pain is common. Up to 10% of the Population has been estimated to suffer from chronic pain and up to 5% of the female population has been estimated to suffer from widespread, chronic pain and tenderness, thus fulfilling American College of Rheumatology (ACR) criteria for classification of fibromyalgia syndrome (FMS). FMS is characterized by the presence of both allodynia and hyperalgesia. FMS is also characterized by disturbances of the autonomic nervous system such as orthostatic intolerance, postural tachycardia etc. The effect of these conditions during gestation and post partum periods is not well known.

Parturition is a complex process which involves multiple endocrine and physiological changes within a short period of time. Severe pain is an important attribute of this natural process. The purpose of the current study is to evaluate the impact of chronic central pain on the process of parturition. Our hypothesis is, that women demonstrating signs, symptoms and a history of central pain, before the onset of active labor, will differ from women not demonstrating such traits; these women may require earlier higher does of analgesia, and may demonstrate increased hemodynamic lability during labor and delivery.

DETAILED DESCRIPTION:
Chronic pain is common. Up to 10% of the Population has been estimated to suffer from chronic pain and up to 5% of the female population has been estimated to suffer from widespread, chronic pain and tenderness, thus fulfilling American College of Rheumatology (ACR) criteria for classification of fibromyalgia syndrome (FMS)(1;2). FMS is considered to represent a prototype of chronic pain which is mediated by the central nervous system, i.e. a condition in which chronic pain is the result of augmented pain processing (and diminished pain - inhibition) within the Central Nercous System (CNS) circuitry (3). Clinical characteristics which are suggestive of the presence of central, versus peripheral (nociceptive) or neuropathic pain, are a lifetime history of pain conditions, a diffuse, non- anatomical distribution of pain, a family history of chronic pain and the co-existence of additional "functional" symptoms such as chronic fatigue, disturbed sleep, irritable bowel etc.

The current paradigms accepted for the pathogenesis of central pain involve an imbalance of multiple neurotransmitters in the CNS, some inhibitory (e.g. serotonin, norepinephrine) others facilitatory (e.g. substance P) which govern the process of spinal pain transmission. Additional processing takes place at higher centers, such as the amygdala and thalamus (4).

FMS is characterized by the presence of both allodynia and hyperalgesia. In addition, medications which have been shown to be effective in FMS and similar conditions are different from those effective in acute pain or in other chronic pain conditions not characterized as central (e.g. malignancy - associated pain). Thus, opioids and Non Steroidal Anti-Inflammatory Drugs (NSAIDS) are relatively ineffective for the treatment of central pain (the former may even cause paradoxical hyperalgesia) (5) while medications which increase levels of norepinephrine and serotonin (NSRIs) are often effective. FMS is also characterized by disturbances of the autonomic nervous system such as orthostatic intolerance, postural tachycardia etc.(6) The effect of these conditions during gestation and post partum periods is not well known.

Parturition is a complex process which involves multiple endocrine and physiological changes within a short period of time. Severe pain is an important attribute of this natural process. The processes of labor, delivery and also the peripartum period are characterized by acute shifts in volume, loss of blood and additional forms of physiological stress and emotional distress.

The purpose of the current study is to evaluate the impact of chronic central pain on the process of parturition. Our hypothesis is, that women demonstrating signs, symptoms and a history of central pain, before the onset of active labor, will differ from women not demonstrating such traits; these women may require earlier higher does of analgesia, and may demonstrate increased hemodynamic lability during labor and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, week 39-41
* Ability to give written informed consent

Exclusion Criteria:

* Age under 18
* High risk pregnancy
* Not able to give written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted as an open label, observational research. The setting of the study is the Obstetric ER of the Lis Maternity Hospital, Tel Aviv sourasky medical center.
  Participants in the study will be pregnant women attending the obstetric ER for routine term followup. This evaluation is generally conducted at week 39-41 of pregnancy. The current study will focus on women attending a regular followup, not considered to be at high risk.
  All participants will be requested to sign written informed consent on recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Patient Controlled Analgesia (PCA) use during delivery | up to 3 days after delivery
  Use of anagesics (i.e. PCA) during and after delivery will be documented and compared with results of evaluation performed before delivery regarding tenderness, symptoms of fibromyalgia etc/

SECONDARY OUTCOMES:
Patient report of pain intensity during delivery | up to 3 days after delivery
  Information will be collected regarding pain levels during delivery, regarding hemodynamic changes during delivery, regarding the mode of delivery as well as standard neonatal data (APGAR score etc)
Blood pressure and pulse recordings | During labor
  Standard clinical recording of hemodynamic measurments during labor
Mode of delivery | During labor
  Recording of mode of delivery, need for cessarian section etc

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Ceter, Tel Aviv, Israel, Israel

REFERENCES:
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Ablin K, Clauw DJ. From fibrositis to functional somatic syndromes to a bell-shaped curve of pain and sensory sensitivity: evolution of a clinical construct. Rheum Dis Clin North Am. 2009 May;35(2):233-51. doi: 10.1016/j.rdc.2009.06.006. PMID 19647139
- [Background] Eisenberg E, McNicol ED, Carr DB. Efficacy and safety of opioid agonists in the treatment of neuropathic pain of nonmalignant origin: systematic review and meta-analysis of randomized controlled trials. JAMA. 2005 Jun 22;293(24):3043-52. doi: 10.1001/jama.293.24.3043. PMID 15972567
- [Background] Cohen H, Neumann L, Shore M, Amir M, Cassuto Y, Buskila D. Autonomic dysfunction in patients with fibromyalgia: application of power spectral analysis of heart rate variability. Semin Arthritis Rheum. 2000 Feb;29(4):217-27. doi: 10.1016/s0049-0172(00)80010-4. PMID 10707990